CLINICAL TRIAL: NCT00055640
Title: Molecular Risk Guided Treatment Of Diffuse Large B-Cell Non-Hodgkin's Lymphoma
Brief Title: Molecular Risk Assessment in Planning Treatment for Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Omer N. Koc, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1402; P30CA043703 (NIH); CWRU-060244; CWRU-1402
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Lymphoma
Keywords: stage I adult diffuse large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; Microarray Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: rituximab — Rituximab IV over 3-6 hours.Treatment repeats every 21 days for 3-8 courses.
Drug: cyclophosphamide — Cyclophosphamide IV over 30 minutes. Treatment repeats every 21 days for 3-8 courses.
Drug: doxorubicin hydrochloride — Doxorubicin IV over 5 minutes. Treatment repeats every 21 days for 3-8 courses.
Drug: prednisone — Oral prednisone on days 1-5. Treatment repeats every 21 days for 3-8 courses.
Drug: vincristine sulfate — Vincristine IV over 5 minutes on day 1. Treatment repeats every 21 days for 3-8 courses.
Genetic: microarray analysis — genetic testing

SUMMARY:
RATIONALE: Analyzing genes that are present in cancer cells may be useful as a method for predicting the response of non-Hodgkin's lymphoma to cancer treatment. Imaging procedures such as positron emission tomography (PET) scans may improve the ability to measure how well cancer has responded to treatment.

PURPOSE: This phase II trial is studying molecular risk assessment to see how well it works in predicting response to therapy in patients who are receiving treatment for non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether molecular risk assessment can identify groups of patients with diffuse large B-cell non-Hodgkin's lymphoma (NHL) who will demonstrate at least 50% difference in early response rates to treatment as determined by positron-emission tomography (PET) imaging.
* Determine, by PET imaging, the response rate of patients treated with cyclophosphamide, doxorubicin, vincristine, prednisone, and rituximab.
* Determine whether early response rates can be predicted by gene expression profiles at diagnosis in these patients.
* Compare gene expression profiles of patients with refractory or relapsed large cell NHL with profiles of the disease at diagnosis.
* Determine relapse-free and overall survival rates of these patients.
* Determine the feasibility of a new NHL treatment algorithm based on prognostic index and molecular risk, and early response assessment by PET imaging.

OUTLINE: Molecular risk assessment is performed using lymph node tissue from initial diagnosis to test for "activated" genes before starting treatment.

Patients receive rituximab IV over 3-6 hours, cyclophosphamide IV over 30 minutes, doxorubicin IV over 5 minutes, and vincristine IV over 5 minutes on day 1 and oral prednisone on days 1-5. Treatment repeats every 21 days for 3-8 courses. Patients undergo whole-body positron-emission tomography (PET) scanning at baseline and after course 3 to determine response. Results from the genetic testing and PET scans are used to determine further treatment recommendations.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 36-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diffuse large B-cell non-Hodgkin's lymphoma
* CD20 and/or CD19 positive by immunohistochemistry or flow cytometry
* Disease evaluable by positron-emission tomography scan
* Diagnostic tissue (either frozen or fresh unfixed) available for molecular testing or willing to undergo a repeat procedure to obtain such tissue
* No CNS involvement by lymphoma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 3 mg/dL

Renal

* Creatinine no greater than 3 mg/dL

Cardiovascular

* LVEF at least 40%

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No significant organ dysfunction that would preclude study chemotherapy
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy
* No prior biological response modifier therapy

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy
* No prior radioimmunotherapy

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2002-10; Primary Completion 2005-04 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Molecular risk assessment to see how well it works in predicting response to therapy in patients who are receiving treatment for non-Hodgkin's lymphoma. | Results from the genetic testing and PET scans at baseline and after course 3 to determine response.

CONTACTS AND LOCATIONS:
Overall Officials: Omer N. Koc, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States